CLINICAL TRIAL: NCT06415474
Title: Evolution of the Lymphocyte Phenotype in Patients with Infection in Intensive Care Unit
Acronym: REAPHEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29BRC23.0109
Record Dates: First submitted 2024-04-26; First posted 2024-05-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Patients Undergoing Esophagectomy; Patients with Severe Polytrauma; Patients with Severe Neurological Lesion; Patients with Abdominal Infection

STUDY DESIGN:
Intervention Model Description: For all patients, lymphocyte phenotyping will be performed on biological samples taken on D0, D7 and the day of discharge. In case of infection, phenotyping will also be performed on the day of infection diagnosis and on the day corresponding to half the duration of antibiotic therapy.
  For phenotyping, only 1.5 mL (0.5 mL per analysis) will be used (if no infection). In case of infection, an additional 1mL will be collected (0.5mL on the day of inclusion diagnosis and 0.5 mL on the day corresponding to half the duration of antibiotic therapy). Blood is collected during sampling, which takes place several times a day as part of the standard management of these patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phenotyping arm (Other): There is only one arm in the study. All patients (i.e. our 4 target populations) will undergo the same phenotyping procedure.
  Interventions: Procedure: Lymphocyte Phenotyping Procedure

INTERVENTIONS:
Procedure: Lymphocyte Phenotyping Procedure — For all patients, lymphocyte phenotyping will be performed on biological samples taken on D0, D7 and the day of discharge. In case of infection, phenotyping will also be performed on the day of infection diagnosis and on the day corresponding to half the duration of antibiotic therapy.
  For phenotyping, only 1.5 mL will be used. In case of infection, an additional 1mL will be collected (0.5mL on the day of inclusion diagnosis and 0.5 mL on the day corresponding to half the duration of antibiotic therapy). Blood is collected during sampling, which takes place several times a day as part of the standard management of these patients.
  It is important to note that phenotyping is not routinely performed as part of routine care. An additional tube is therefore taken specifically for this analysis, but this is done without the need for an additional puncture.

SUMMARY:
Patients admitted for polytrauma, severe neurological injury, post-operative monitoring or sepsis/septic shock present with significant inflammation, leading to immunoparalysis, which is responsible for infection, particularly prolonged infection. A study of their lymphocyte phenotype over time could help explore the phenomenon of immunoparalysis.

ELIGIBILITY:
Inclusion criteria:

* Postoperative esophagectomy surveillance within the last 24 hours.
* Patients with intra-abdominal infection
* Neurological patients with intubation planned for more than 24 hours (subarachnoid hemorrhage with coma, severe head trauma, ischemic or hemorrhagic stroke with coma).
* Polytrauma with intubation planned for more than 24 hours
* Patient aged 18 and over
* Patient with social security coverage

Non-inclusion criteria :

* Hereditary immune deficiency HIV-AIDS
* Malignant hemopathies
* Immunosuppressive treatment other than corticosteroid therapy or chemotherapy
* Patient under legal protection
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2026-10-03 (Estimated); Study Completion 2026-11-03 (Estimated)

PRIMARY OUTCOMES:
Lymphocytes numbers variation | Day 0
  - Numbers of various lymphocytes (LT, LB, NK and their subclasses) at D0 according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes numbers variation | Day 7
  - Numbers of various lymphocytes (LT, LB, NK and their subclasses) at D7 according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes numbers variation | Immediately upon prescribed discharge date
  - Numbers of various lymphocytes (LT, LB, NK and their subclasses) at discharge according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes numbers variation | Immediately after diagnosis of infection
  - Numbers of various lymphocytes (LT, LB, NK and their subclasses) at diagnosis of infection according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes numbers variation | At the midpoint of the prescribed antibiotic course
  - Numbers of various lymphocytes (LT, LB, NK and their subclasses) at half duration of infection's treatment according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes percentages variation | Day 0
  - Percentage rate of various lymphocytes (LT, LB, NK and their subclasses) at D0 according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes percentages variation | Day 7
  - Percentage rate of various lymphocytes (LT, LB, NK and their subclasses) at D7 according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes percentages variation | Immediately upon prescribed discharge date
  - Percentage rate of various lymphocytes (LT, LB, NK and their subclasses) at discharge according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes percentages variation | Immediately after diagnosis of infection
  - Percentage rate of various lymphocytes (LT, LB, NK and their subclasses) at day of diagnosis according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)
Lymphocytes percentages variation | At the midpoint of the prescribed antibiotic course
  - Percentage rate of various lymphocytes (LT, LB, NK and their subclasses) at half duration of infection's treatment according to reason for admission (postoperative vs sepsis/septic shock vs polytrauma vs neurological injury)

SECONDARY OUTCOMES:
Lymphocytes percentages variation in case of infection | Day 0
  Percentage rate in various lymphocytes (LT, LB, NK and their subclasses) at D0
Lymphocytes percentages variation in case of infection | At the onset of symptoms of infection
  Percentage rate in various lymphocytes (LT, LB, NK and their subclasses) at onset of infection
Lymphocytes percentages variation in case of infection | Immediately following resolution of infection
  Percentage rate in various lymphocytes (LT, LB, NK and their subclasses) at resolution of infection
Lymphocytes numbers variation in case of infection | Day 0
  Numbers rate in various lymphocytes (LT, LB, NK and their subclasses) at D0
Lymphocytes numbers variation in case of infection | Immediately after diagnosis of infection
  Numbers rate in various lymphocytes (LT, LB, NK and their subclasses) at onset of infection
Lymphocytes numbers variation in case of infection | Immediately following resolution of infection
  Numbers rate in various lymphocytes (LT, LB, NK and their subclasses) at resolution of infection

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided